CLINICAL TRIAL: NCT02258425
Title: Homeless Female Offenders Returning to the Community: Improving Hopeful Futures
Brief Title: Homeless Female Offenders Returning to the Community
Acronym: FEM-CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Adeline Nyamathi, PhD, Distinguished Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1R34DA035409 (NIH)
Record Dates: First submitted 2014-10-02; First posted 2014-10-07 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Drug Addiction
Keywords: Homeless Women; Parolees; Probationers; Community Drug Treatment; Recidivism
MeSH Terms: conditions — Substance-Related Disorders; Recidivism | interventions — Health Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FEM-CARE (Experimental): Six specialized nurse case managed and health education sessions and coach-facilitated mentoring
  Interventions: Behavioral: FEM-CARE
- Health Promotion (Active Comparator): One brief basic health education session and coach-facilitated mentoring
  Interventions: Behavioral: Health Promotion

INTERVENTIONS:
Behavioral: FEM-CARE
  Arms: FEM-CARE
Behavioral: Health Promotion
  Arms: Health Promotion

SUMMARY:
In Phase I of this R34, the team from the University of California Los Angeles, San Francisco, and Irvine researchers plan to utilize the successful community participatory approaches to refine a gender-sensitive criminogenic needs -focused intervention program, Female Ex-Offender Mentoring in Care (FEM-CARE), with the help of a community advisory board, composed of homeless female offenders (HFOs) and addiction staff; and finalize strategies which will be validated by focus group sessions with the HFOs. In Phase 2, the research team will randomize 130 HFOs participating in one of two residential drug treatment programs to assess the impact of the FEM-CARE or a Health Promotion control program on reduction of drug and alcohol use and recidivism. This study is based upon our team's history of promoting theoretically-based, culturally sensitive nurse-led interventions that are enriched with criminal justice theoretical perspectives, and have resulted in significant reductions in drug and alcohol use among homeless persons, many of whom have had a history of incarceration.

Specifically, the study aims are:

AIM 1) Guided by a Community Advisory Board (CAB) made up of HFOs and addiction staff, further conceptualize our community-based program, Female Ex-Offender Mentoring in Care (FEM-CARE), to address the needs and risks of HFOs enrolled in RDT programs, and then refine the program in focus group discussions with 12 HFOs.

AIM 2) Conduct a pilot RCT to assess the impact of the FEM-CARE program for 65 HFOs at six-month follow-up compared with 65 HFOs receiving a control Health Promotion (HP) program, in terms of a) self-reported and/or objective measures of drug and alcohol use; and b) prevalence of recidivism and number of days to first reincarceration.

Hypothesis 2a: HFOs in the FEM-CARE program will have less drug and alcohol use at six months than HFOs in the HP control program.

Hypothesis 2b: FEM-CARE HFOs will have a lower prevalence of recidivism by six months and greater number of days to first reincarceration than HP control HFOs.

DETAILED DESCRIPTION:
In the last decade, the numbers of incarcerated females has tripled, making women the most rapidly growing group of offenders in the United States. When compared to incarcerated males, female offenders have a higher rate of being sentenced for drug crimes; moreover, they are often injection drug users (IDUs), have sexual partners who are IDUs, and are often forced into the sex trade for survival. As many as 50% of female offenders report physical and/or sexual abuse; further, traumatic abuse, chronic emotional distress, and internalized stigma resulting from being a felon and a drug-user, have a profound effect on the women's self-esteem, leading to feelings of hopelessness and depression, delayed recovery and reintegration, increased risky behaviors, and health concerns. Not surprisingly, women who have been incarcerated are nearly twice as likely to experience mental illness compared with non-offending women; further, 44% recidivate within a year due to possession of a controlled substance. In particular, among homeless female offenders (HFOs), both parolees and probationers report ongoing challenges for successful re-entry. These include unstable housing, disorganized lives, unemployment, and limited access to health and social services. While the Los Angeles County Department of Probation has provided guidance for successful programs in its California Blueprint Master Plan for Female Offenders, the suggested strategies of enhancing empowerment, positive coping, and job skills, and providing peer-mentored approaches have not yet been implemented or evaluated. In Phase I of this R34, our team of University of California Los Angeles, San Francisco, and Irvine researchers plan to utilize our successful community participatory approaches to refine a gender-sensitive criminogenic needs -focused intervention program, Female Ex-Offender Mentoring in Care (FEM-CARE), with the help of a community advisory board, composed of HFOs and addiction staff; and finalize strategies which will be validated by focus group sessions with HFOs. In Phase 2, we will randomize 130 HFOs participating in one of two residential drug treatment programs to assess the impact of the FEM-CARE or a Health Promotion control program on reduction of drug and alcohol use and recidivism. This study is based upon our team's history of promoting theoretically-based, culturally sensitive nurse-led interventions that are enriched with criminal justice theoretical perspectives, and have resulted in significant reductions in drug and alcohol use among homeless persons, many of whom have had a history of incarceration. Our most recent successes in engaging male parolees in nurse-supported peer mentorship, our team's expertise in enhancing stigma reduction among vulnerable women, and our criminal justice experts have informed this study. Finally, recent formative research with HFOs has revealed a desire for peer role models to support and enhance knowledge of and access to healthcare, promote positive coping, stable housing, and job skills, and to reduce stigma and depressed mood; all of these factors can result in novel programs designed to prevent drug and alcohol use and reduce recidivism. This foundation and strong community support garnered has led to the design of our proposed intervention program.

ELIGIBILITY:
Inclusion Criteria:

* female parolees or probationers enrolled in a six-month program at one of two residential treatment (RDT) programs,
* convicted for a drug crime, and
* reported homeless on their RDT entry form

Exclusion Criteria:

* female parolees or probationers not currently enrolled in a six-month program at one of two residential treatment (RDT) programs,
* not recently convicted for a drug crime, and
* not reported homeless on their RDT entry form

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | 3 years
  Reduction in drug and alcohol use

SECONDARY OUTCOMES:
Secondary Outcome Measure | 3 years
  Number of visits to health care or social service providers

CONTACTS AND LOCATIONS:
Overall Officials: Adeline Nyamathi, PhD, Principal Investigator — UCLA/UCI
Locations (1):
- Amistad de Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nyamathi AM, Srivastava N, Salem BE, Wall S, Kwon J, Ekstrand M, Hall E, Turner SF, Faucette M. Female Ex-Offender Perspectives on Drug Initiation, Relapse, and Desire to Remain Drug Free. J Forensic Nurs. 2016 Apr-Jun;12(2):81-90. doi: 10.1097/JFN.0000000000000110. PMID 27195929
- [Background] Nyamathi AM, Salem BE, Hall E, Oleskowicz T, Ekstrand M, Yadav K, Toyama J, Turner S, Faucette M. Violent Crime in the Lives of Homeless Female Ex-Offenders. Issues Ment Health Nurs. 2017 Feb;38(2):122-131. doi: 10.1080/01612840.2016.1253807. Epub 2017 Feb 2. PMID 28152325
- [Derived] Nyamathi AM, Shin SS, Smeltzer J, Salem BE, Yadav K, Ekstrand ML, Turner SF, Faucette M. Achieving Drug and Alcohol Abstinence Among Recently Incarcerated Homeless Women: A Randomized Controlled Trial Comparing Dialectical Behavioral Therapy-Case Management With a Health Promotion Program. Nurs Res. 2017 Nov/Dec;66(6):432-441. doi: 10.1097/NNR.0000000000000249. PMID 29095374